CLINICAL TRIAL: NCT05395910
Title: Phase 1 Study of Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) and Electrostatic PIPAC (ePIPAC) With Paclitaxel for Peritoneal Carcinomatosis - PIPAC2 Study
Brief Title: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) and Electrostatic PIPAC (ePIPAC) With Paclitaxel In Patients With Peritoneal Carcinomatosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSRB 2020/01447
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Peritoneal Carcinomatosis
Keywords: Gastric Cancer; Oesophageal Cancer; Bilio-pancreatic tract Cancer; Gynaecological Cancer; Colorectal Cancers; Unresectable Peritoneal Carcinomatosis; Pressurized intraperitoneal aerosol chemotherapy; Electrostatic precipitation pressurized intraperitoneal aerosol chemotherapy; Paclitaxel
MeSH Terms: conditions — Peritoneal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIPAC Paclitaxel (Experimental): 3 patients will be allocated to PIPAC arm at Paclitaxel 15mg/m2. If there is 1 dose limiting toxicity (DLT), an additional 3 patients will be allocated to PIPAC arm at 15mg/m2. If there is 2 - 3 DLT, study had exceeded its Maximum Tolerable Dose (MTD) and we will proceed to stop recruitment.
  Should there be no DLT, recruitment at PIPAC 30mg/m2 and ePIPAC 15mg/m2 will occurs concurrently in an alternating fashion. PIPAC/ePIPAC dose escalation will continue until a MTD has been reached. Should there be no DLT at PIPAC 30mg/m2 and ePIPAC 15mg/m2, recruitment at PIPAC 45mg/m2 and ePIPAC 30mg/m2 will occurs concurrently in an alternating fashion. Finally, should there be no DLT, recruitment at ePIPAC 45mg/m2 will occurs.
  Interventions: Drug: Paclitaxel
- ePIPAC Paclitaxel (Experimental): Should there be no DLT under PIPAC arm at Paclitaxel 15mg/m2, recruitment at ePIPAC 15mg/m2 and PIPAC 30mg/m2 will occurs concurrently in an alternating fashion. PIPAC/ePIPAC dose escalation will continue until a MTD has been reached. Should there be no DLT at PIPAC 30mg/m2 and ePIPAC 15mg/m2, recruitment at PIPAC 45mg/m2 and ePIPAC 30mg/m2 will occurs concurrently in an alternating fashion. Finally, should there be no DLT, recruitment at ePIPAC 45mg/m2 will occurs.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — This is a prospective, two armed phase I trial in a 3 + 3 dose escalation evaluating the safety and tolerability of PIPAC/ePIPAC using paclitaxel in patients with peritoneal carcinomatosis.

SUMMARY:
Peritoneal carcinomatosis (PC) is a miserable disease with poor treatment outcome. Intraperitoneal administration of anticancer drugs enables an extremely high concentration of drugs to directly contact the target cancer lesions in the peritoneal cavity. However, its effectiveness is limited by the intraperitoneal distribution and penetration of the drug. Pressurized intraperitoneal aerosol chemotherapy (PIPAC) is an innovative intraperitoneal chemotherapy concept that enhances efficacy by taking advantage of the physical properties of gas and pressure. Electrostatic precipitation pressurized intraperitoneal aerosol chemotherapy (ePIPAC) may further enhance these benefits.

This research study serves to determine the safety profile and tolerability of PIPAC/ePIPAC with paclitaxel. It will determine the maximal tolerated dose (MTD) and evaluate the safety and tolerability, and pharmacokinetics of PIPAC/ePIPAC paclitaxel in pre-treated patients with peritoneal carcinomatosis (PC). It may offer a novel and effective option of treatment for patients with PC, who, at present have limited options involving the use of systemic chemotherapy and who suffer from poor life expectancy and poor quality of life.

DETAILED DESCRIPTION:
In patients with histologically proven unresectable or recurrent gastric cancer limited to the peritoneum, the combination of intraperitoneal (IP) paclitaxel with systemic chemotherapy reported a one-year survival rate of 78%. However, the effectiveness of IP chemotherapy may be limited by its distribution, tissue penetration and associated catheter-related complications.

Pressurized Intra-Peritoneal Aerosol Chemotherapy (PIPAC) is a novel drug delivery technique for PC taking advantage of physical laws (gaseous nature, hydrostatic pressure) with superior pharmacological properties (homogeneous distribution, deeper tissue penetration). It is applied through laparoscopy and is minimally invasive. Adding electrostatic loading (ePIPAC) as an adjunct would further improve the pharmacological properties of PIPAC since it should induce precipitation of the aerosolized drug, increasing the ratio between the dose applied and the dose in the target tissue.

Systemic toxicity is significantly reduced due to the peritoneum/blood barrier and the low dose applied (about 20% of the usual systemic dose). A systematic review highlighted that PIPAC combines the benefits of a minimally invasive approach with pharmacokinetic advantages of intraperitoneal administration and pressurized vaporization. It concluded that PIPAC is feasible, safe, and warrants further prospective studies. PIPAC may be combined with systemic palliative chemotherapy with minimal additional organ toxicity. This method of treatment avoids the morbidity and mortality of HIPEC. PIPAC has been shown in pre-clinical studies to be potentially more efficacious than catheter-based IP-chemotherapy due to better drug distribution and penetration. In clinical use, PIPAC can be repeated at intervals of 6 weeks to 3 months. This allows repeated objective assessment of therapy effect over time.

To date, PIPAC has only been utilized to administer Oxaliplatin or a combination of Doxorubicin/Cisplatin. Paclitaxel is an approved drug for systemic chemotherapy for several cancers, and also has well-documented intraperitoneal use for ovarian cancer and gastric cancer. It is a hydrophobic, high molecular weight compound resulting in low absorption through the lymphatic system after IP administration with a much higher peritoneal to plasma peak concentration and AUC ratios (>1000 versus 25 and >1000 versus 16 respectively). As such, IP Paclitaxel may be potentially more efficacious with less systemic toxicity than IP Oxaliplatin. However, no clinical data exists in the published literature for PIPAC/ePIPAC paclitaxel.

This proposed prospective study is the first clinical study of PIPAC/ePIPAC with Paclitaxel. It will determine the maximal tolerated dose (MTD) and evaluate the safety and tolerability, and pharmacokinetics of PIPAC/ePIPAC paclitaxel in pre-treated patients with PC. Peritoneal biopsies will be collected prior to and after PIPAC/ePIPAC to assess tissue drug concentration and depth of drug penetration. Collection of biospecimens including peritoneal tissue, peritoneal fluid and blood will be used for correlative studies including paclitaxel resistance analysis and development of cancer modelling platforms. For the individual patient, repeated biopsies and molecular profiling may also facilitate individualized therapy. For medical research, PIPAC/ePIPAC may deliver measurable progress in 3-5 years because the assessment interval is short (6 weeks) in this disease with rapid progression (6-12 months to death).

This study will determine the safety dose range of PIPAC/ePIPAC paclitaxel. This will allow us to design a phase II trial to evaluate clinical efficacy. On a larger scale, the success of this PIPAC/ePIPAC trial would add a valuable treatment option to our arsenal in the treatment of PC.

ELIGIBILITY:
Inclusion Criteria:

* All solid cancer patients with peritoneal metastasis on peritoneal cytology/histology.
* Patients who refuse, are unable to tolerate, or have completed at least 1st line systemic chemotherapy
* Patients who have completed chemotherapy/targeted therapy > 21 days or at least 5 half-lives (whichever is longer) prior to PIPAC/ePIPAC
* Patients must have recovered (≤ grade 1) from all reversible treatment toxicity from prior chemotherapy, radiotherapy or surgery.
* Age ≥21 years
* Eastern Cooperative Oncology Group performance status 0-2
* Adequate bone marrow function (neutrophil count ≥1500/mm3, hemoglobin ≥8.0 g/dl and platelet count ≥100 000/mm3)
* Adequate liver function (bilirubin ≤ 1.5x ULN (upper limit normal) and AST/ALT ≤3x ULN or ≤5x ULN in the presence of liver metastases)
* Adequate renal function (serum creatinine ≤1.5x ULN)
* Expected survival >3 months
* Able to understand and the willingness to sign a written informed consent document
* The effects of proposed regimen on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because antitumor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Patients with treated skin cancer besides melanoma may be included.

Exclusion Criteria:

* Predominant extra-peritoneal metastases at the discretion of the study team after discussion at the multidisciplinary tumor board
* Patients with clinical or radiological evidence of hollow viscera perforation or impending perforation, including but not limited to gastric, small bowel, colon, gallbladder. Decision will be made at the discretion of the study team in consultation with multidisciplinary tumour board or with necessary specialists
* Good response to systemic chemotherapy based on RECIST guidelines version 1.1 with complete or partial response to systemic chemotherapy
* Known allergy to paclitaxel
* Previous malignancy unrelated to current peritoneal carcinomatosis diagnosed in the last 2 years
* Patients with reproductive potential who refuse to use an adequate means of contraception (including male patients)
* Significant disease or conditions which, in the investigator's opinion, would exclude patient from the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating female
* Patients with bowel obstruction, total dependence on parenteral nutrition, or who are undergoing gastrointestinal resection in the same setting

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tolerability of PIPAC /ePIPAC with Paclitaxel by monitoring dose limiting toxicities | 1 - 2 years
  Dose limiting toxicities are monitored to evaluate the tolerability of PIPAC /ePIPAC
Safety Profile of PIPAC/ePIPAC with Paclitaxel by monitoring adverse events | 1 - 2 years
  Adverse events are monitored to evaluate the safety profile of PIPAC/ePIPAC

SECONDARY OUTCOMES:
Clinical response of PIPAC/ePIPAC with Paclitaxel according to Peritoneal Cancer Index (PCI) | 1 - 2 years
  Peritoneal Cancer Index (PCI) is used to measure Clinical response of PIPAC/ePIPAC with Paclitaxel
Pathological response of PIPAC/ePIPAC with Paclitaxel according to Peritoneal Regression Grade Scoring (PRGS) System | 1 - 2 years
  Peritoneal Regression Grade Scoring (PRGS) System is used to measure Pathological response of PIPAC/ePIPAC
Maximum concentration (Cmax) of Paclitaxel administered via PIPAC/ePIPAC using blood drawn from patient. | Pre-dose; 30 and 45 minutes; and 1, 2, 4, 8, 24, 30, 48 hour
Half-life (t1/2) of Paclitaxel administered via PIPAC/ePIPAC using blood drawn from patient | Pre-dose; 30 and 45 minutes; and 1, 2, 4, 8, 24, 30, 48 hour
Area under the curve (AUC) of Paclitaxel administered via PIPAC/ePIPAC using blood drawn from patient. | Pre-dose; 30 and 45 minutes; and 1, 2, 4, 8, 24, 30, 48 hour

CONTACTS AND LOCATIONS:
Overall Officials: Bok Yan Jimmy So, MBChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishigami H, Kitayama J, Kaisaki S, Hidemura A, Kato M, Otani K, Kamei T, Soma D, Miyato H, Yamashita H, Nagawa H. Phase II study of weekly intravenous and intraperitoneal paclitaxel combined with S-1 for advanced gastric cancer with peritoneal metastasis. Ann Oncol. 2010 Jan;21(1):67-70. doi: 10.1093/annonc/mdp260. Epub 2009 Jul 15. PMID 19605503
- [Background] Kobayashi D, Kodera Y. Intraperitoneal chemotherapy for gastric cancer with peritoneal metastasis. Gastric Cancer. 2017 Mar;20(Suppl 1):111-121. doi: 10.1007/s10120-016-0662-9. Epub 2016 Nov 1. PMID 27803990
- [Background] Solass W, Hetzel A, Nadiradze G, Sagynaliev E, Reymond MA. Description of a novel approach for intraperitoneal drug delivery and the related device. Surg Endosc. 2012 Jul;26(7):1849-55. doi: 10.1007/s00464-012-2148-0. Epub 2012 May 12. PMID 22580869
- [Background] Solass W, Herbette A, Schwarz T, Hetzel A, Sun JS, Dutreix M, Reymond MA. Therapeutic approach of human peritoneal carcinomatosis with Dbait in combination with capnoperitoneum: proof of concept. Surg Endosc. 2012 Mar;26(3):847-52. doi: 10.1007/s00464-011-1964-y. Epub 2011 Nov 1. PMID 22042585
- [Background] Grass F, Vuagniaux A, Teixeira-Farinha H, Lehmann K, Demartines N, Hubner M. Systematic review of pressurized intraperitoneal aerosol chemotherapy for the treatment of advanced peritoneal carcinomatosis. Br J Surg. 2017 May;104(6):669-678. doi: 10.1002/bjs.10521. PMID 28407227
- [Background] Reymond M, Demtroeder C, Solass W, Winnekendonk G, Tempfer C. Electrostatic precipitation Pressurized IntraPeritoneal Aerosol Chemotherapy (ePIPAC): first in-human application. Pleura Peritoneum. 2016 Jun 1;1(2):109-116. doi: 10.1515/pp-2016-0005. Epub 2016 Apr 29. PMID 30911614
- [Background] Ishigami H, Fujiwara Y, Fukushima R, Nashimoto A, Yabusaki H, Imano M, Imamoto H, Kodera Y, Uenosono Y, Amagai K, Kadowaki S, Miwa H, Yamaguchi H, Yamaguchi T, Miyaji T, Kitayama J. Phase III Trial Comparing Intraperitoneal and Intravenous Paclitaxel Plus S-1 Versus Cisplatin Plus S-1 in Patients With Gastric Cancer With Peritoneal Metastasis: PHOENIX-GC Trial. J Clin Oncol. 2018 Jul 1;36(19):1922-1929. doi: 10.1200/JCO.2018.77.8613. Epub 2018 May 10. PMID 29746229
- [Background] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Background] Chan DY, Syn NL, Yap R, Phua JN, Soh TI, Chee CE, Nga ME, Shabbir A, So JB, Yong WP. Conversion Surgery Post-Intraperitoneal Paclitaxel and Systemic Chemotherapy for Gastric Cancer Carcinomatosis Peritonei. Are We Ready? J Gastrointest Surg. 2017 Mar;21(3):425-433. doi: 10.1007/s11605-016-3336-3. Epub 2016 Dec 15. PMID 27981493
- [Background] Kono K, Yong WP, Okayama H, Shabbir A, Momma T, Ohki S, Takenoshita S, So J. Intraperitoneal chemotherapy for gastric cancer with peritoneal disease: experience from Singapore and Japan. Gastric Cancer. 2017 Mar;20(Suppl 1):122-127. doi: 10.1007/s10120-016-0660-y. Epub 2016 Oct 20. PMID 27766496